CLINICAL TRIAL: NCT05828810
Title: CLinical Evaluation of ANtiseptic Skin Preparation in Revision Total Joint Arthroplasty of the Hip and Knee - A Vanguard Randomized Controlled Registry Trial (CLEAN Joint Trial)
Brief Title: CLinical Evaluation of ANtiseptic Skin Preparation in Revision Total Joint Arthroplasty of the Hip and Knee
Acronym: CLEANJoint
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4000
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-07

CONDITIONS: Revision Total Hip Arthroplasty (RTHA); Revision Total Knee Arthroplasty
Keywords: prosthetic joint infection; registry-based RCT; PJI
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: This is a multicentre, pragmatic, open label, 2-arm parallel-group Vanguard feasibility RCT.
Masking Description: Data analysts will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine gluconate-alcohol solution (Active Comparator): Chlorhexidine gluconate-alcohol solution is a type of solution that has antiseptic properties, which means it helps to eliminate harmful bacteria on the skin at the time of surgery, and therefore, reduce the risk of infection.
  Interventions: Procedure: Chlorhexidne Gluconate-Alcohol Skin Preparation
- Povidone-iodine solution (Active Comparator): Povidone-iodine solution is a type of solution that has antiseptic properties, which means it helps to eliminate harmful bacteria on the skin at the time of surgery, and therefore, reduce the risk of infection.
  Interventions: Procedure: Poviodine-iodine Skin Preparation

INTERVENTIONS:
Procedure: Chlorhexidne Gluconate-Alcohol Skin Preparation — Participants will undergo skin antisepsis with 4% chlorhexidine gluconate pre-wash, followed by 2% chlorhexidine gluconate with 70% isopropyl alcohol skin preparation.
  The surgical field to be sterilized will be at the discretion of the surgical team, but typically includes the distal torso to ankle for patients undergoing hip arthroplasty and proximal thigh to ankle for patients undergoing knee arthroplasty.
  Pre-wash of the surgical area will be carried out using a wet chlorhexidine surgical scrub brush followed by immediate drying using towels. The definitive preparation will then be carried out using tinted chlorhexidine gluconate-alcohol sponges applied with forceps. The drying time and the minimum number of sponge packs used will comply with the product 'Instructions for Use'. The drapes can be applied as per the surgeon's usual approach and they will be treated according to the institution and surgeon's routine practice for draping and surgical site infection prevention.
  Arms: Chlorhexidine gluconate-alcohol solution
Procedure: Poviodine-iodine Skin Preparation — Participants will undergo skin antisepsis with 7.5% povidone-iodine detergent pre-wash, followed by 10% povidone-iodine skin preparation.
  The surgical field to be sterilized will be at the discretion of the surgical team, but typically includes the distal torso to ankle for patients undergoing hip arthroplasty and proximal thigh to ankle for patients undergoing knee arthroplasty.
  Pre-wash of the surgical area will be carried out using iodine detergent soaked gauze pads followed by immediate drying using towels. The definitive preparation will then be carried out using povidone-iodine soaked gauze pads applied with forceps. The drapes can be applied as per the surgical team's usual approach and they otherwise will be treated according to the institution and surgeon's routine practice for draping and surgical site infection prevention.
  Arms: Povidone-iodine solution

SUMMARY:
The goal of this clinical trial is to compare two types of skin preparation solutions (chlorhexidine gluconate-alcohol solution and povidone-iodine solution) that help eliminate harmful bacteria on the skin at the time of surgery for patients having revision arthroplasty surgery of the hip or knee.

The main outcome of interest for the definitive study is the need for re-operation for a wound complication or an infection of the prosthetic joint within one year after surgery.

For the pilot trial, our main interest is to determine feasibility of a definitive trial. Feasibility outcomes will include: ability to recruit patients, ability to randomize patients, ability to collect complete data, estimate the event rate of our primary outcome, ability to carry out data linkages and determine the accuracy of collected data.

Participants will be contacted at two time points after surgery to complete a 5-minute survey: after 30 days, and after 1 year.

DETAILED DESCRIPTION:
In this trial, participants will be assigned randomly to have their surgical skin site prepared for surgery with either chlorhexidine gluconate-alcohol solution or povidone-iodine solution. These are two types of solutions that have antiseptic properties, which means they help eliminate harmful bacteria on the skin at the time of surgery, and therefore, reduce the risk of infection. Surgeons routinely use either chlorhexidine-based or iodine-based skin preparation solutions at the time of surgery to sterilize the surgical area. However, we don't know which one works best for patients having revision joint replacement surgery. There is a small chance of having an allergic reaction to the chlorhexidine or iodine, but there is no additional risk by participating in this study, as these skin preparation solutions are routinely used in practice.

The main outcome of interest is the need for re-operation for a wound complication or an infection of the prosthetic joint within one year after surgery. Other key outcomes are surgical site infection, mortality, and readmission to hospital. Participants will be contacted 30 days after surgery to complete a survey online, by phone, or in person, which will take approximately 5 minutes to complete. All other outcome data will be collected by phone call, health records, routine hospital monitoring, or electronic registry data at thirty days and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Scheduled to undergo aseptic revision total hip arthroplasty or total knee arthroplasty with exchange of at least one prosthetic component

Exclusion Criteria:

1. Revision for prosthetic joint infection or wound complication
2. Known history of previous prosthetic joint infection in the operative joint
3. Any degree of clinical concern for prosthetic joint infection
4. History of allergy to iodine, chlorhexidine, or alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of accrual | 2 years
  Average number of patients enrolled per month: feasible if 10 or more overall
Ability to deliver intervention the patient is randomized to receive | 2 years
  Feasible if >90% of patients receive correct intervention
Ability to collect complete data from participants | 2 years
  Feasible if >80% of data is collected.
To estimate the aggregate incidence of reoperation for wound complication or PJI at one year | 2 years
  Number of reoperations for wound complication or PJI within one year in each group
Ability to link collected outcome data with ICES datasets | 2 years
  Feasible if linkage is possible in >90% of participants.
Validation of the accuracy of outcome data collected through registries and surveillance programs | 2 years
  a) Valid if >90% agreement (sensitivity, specificity, positive predictive value, negative predictive value) for each outcome (collected at follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Raman Mundi, MD MSc FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Sunnybrook Holland Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No